CLINICAL TRIAL: NCT06078748
Title: The Lifestyle, Exercise, and Diet Trial: A Virtual, Lifestyle Approach to Improve Cognition
Brief Title: The Lifestyle Exercise and Diet Trial (LEAD) 2.0
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Baycrest (Other); Université de Montréal (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Laura Middleton, Assistant Professor, University of Waterloo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 44616
Record Dates: First submitted 2023-06-01; First posted 2023-10-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Subjective Cognitive Decline
MeSH Terms: interventions — Diet; Counseling

STUDY DESIGN:
Intervention Model Description: Factorial randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be masked to intervention group.
  Careful wording will be used to describe the intervention groups to participants as to not disclose whether they are in experimental or control groups. For instance, all participants will be told that they will be receiving different combinations of exercise (stretching/toning is the control for aerobic/resistance exercise) and healthy lifestyle interventions (lifestyle education is control for dietary intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EX + DIET (Experimental): Participants will engage in 3 sessions per week (2 EX, 1 DIET, totaling 4 hours per week), consisting of two virtual group sessions (totaling 3 hours) and one independent session (1 hour) (Table 1). Virtual group sessions will occur in groups of 6-8 participants using the Zoom Healthcare platform (on a computer or tablet).
  Interventions: Behavioral: EX; Behavioral: DIET
- EX + ED (Active Comparator): Participants will engage in 3 sessions per week (2 EX, 1 ED, totaling 4 hours per week), consisting of two virtual group sessions (totaling 3 hours) and one independent session (1 hour) (Table 1). Virtual group sessions will occur in groups of 6-8 participants using the Zoom Healthcare platform (on a computer or tablet).
  Interventions: Behavioral: EX; Behavioral: ED
- STRETCH + DIET (Active Comparator): Participants will engage in 3 sessions per week (2 STRETCH, 1 DIET, totaling 4 hours per week), consisting of two virtual group sessions (totaling 3 hours) and one independent session (1 hour) (Table 1). Virtual group sessions will occur in groups of 6-8 participants using the Zoom Healthcare platform (on a computer or tablet).
  Interventions: Behavioral: DIET; Behavioral: STRETCH
- STRETCH + ED (Placebo Comparator): Participants will engage in 3 sessions per week (2 STRETCH, 1 ED) totaling 4 hours per week), consisting of two virtual group sessions (totaling 3 hours) and one independent session (1 hour) (Table 1). Virtual group sessions will occur in groups of 6-8 participants using the Zoom Healthcare platform (on a computer or tablet)
  Interventions: Behavioral: STRETCH; Behavioral: ED

INTERVENTIONS:
Behavioral: EX — EX involves 2.5hrs of moderate intensity aerobic and resistance exercise per week. EX will be instructed by a clinical exercise physiologist (CEP) or registered kinesiologist (RKIN). The EX session will include a 5min warm-up, 20-30min of moderate intensity aerobic exercise, 20-30min of moderate intensity resistance training, and a 5min cool down. The virtual video session will be pre-recorded, have similar composition, and will be led by the same instructor as the group sessions. This group will also receive the "Adult Strategies Put Into Real World Environments" (ASPIRE) goal strategy training, with goals focused on exercise in order to overcome barriers and increase maintenance of lifestyle changes.
  Other Names: Combined aerobic and resistance exercise
  Arms: EX + DIET; EX + ED
Behavioral: DIET — DIET involves one session per week of diet education delivered by a Registered Dietitian. The DIET session will be 90 minutes during months 1-4, and 30 minutes in months 5 and 6. DIET was developed by our team, emphasizing foods identified as supporting executive function, memory, and other cognitive abilities. This group will also receive the "Adult Strategies Put Into Real World Environments" (ASPIRE) goal strategy training, with goals focused on diet in order to overcome barriers and increase maintenance of lifestyle changes.
  Other Names: Brain-healthy diet education and counseling
  Arms: EX + DIET; STRETCH + DIET
Behavioral: STRETCH — STRETCH sessions will be time/frequency-matched to EX sessions (2.5hrs/week: 1.5hr in virtual group sessions; 1hr virtual video session) to control for social aspects and placebo effects of EX.Each STRETCH session will include a 5min warm-up, 5min of balance exercises, and 50min of stretching. Difficulty will not be progressed. STRETCH sessions will also be led by a CEP/RKIN instructor and video sessions will be pre-recorded by the same instructor.
  Other Names: Stretching and toning exercise
  Arms: STRETCH + DIET; STRETCH + ED
Behavioral: ED — ED sessions designed to be of equal intensity and social engagement to the DIET intervention. Participants will engage in group discussion and receive information on the brain and cognitive processes, the effect of age on cognition, and tips to promote healthy aging. This will include lectures, watching documentaries and participating in various games.
  Other Names: Brain Health Education and Discussion
  Arms: EX + ED; STRETCH + ED

SUMMARY:
The objective of this study is to investigate the feasibility of a virtually-delivered 6-month exercise and nutrition intervention in older adults with executive subjective cognitive decline (SCD). Feasibility will be determined by recruitment, retention, and adherence rates. Preliminary changes in cognition, physical function, and quality of life will be assessed as secondary outcomes. The study will recruit 140 participants aged 65 to 80 who report they feel that their memory or other thinking abilities are declining. Participants will be randomized into one of four study arms receiving different combinations of healthy lifestyle interventions. Assessments will be conducted virtually at baseline, post-intervention (6 months), and follow-up (12 months). All intervention sessions and assessment visits will be conducted online using the Zoom Healthcare platform and participants will log on using their own devices from home.

DETAILED DESCRIPTION:
The study will be a randomized control trial examining the feasibility of a 6-month virtually delivered exercise and nutrition intervention in older adults with executive SCD. The study aims to recruit 140 participants. After initial contact with potential participants, 2 screening visits (up to 45 minutes each) will be conducted to assess eligibility and obtain consent to participate in the study. At the start of the program, after completing the program (6 months), and at follow-up (12 months), assessors will conduct 2 assessments (30-65 min each) using Zoom video conferencing to measure thinking abilities, physical function, and quality of life. Participants will be randomized into one of four 6-month intervention arms (35 individuals per group x 4 groups): 1) EX + DIET: aerobic and resistance exercise (EX) with healthy diet counseling (DIET), 2) EX + ED: aerobic and resistance exercise (EX) with education on healthy lifestyle related to brain health (ED), 3) STRETCH + DIET: stretching and toning exercises (STRETCH) with healthy diet counseling (DIET), 4) STRETCH + ED: stretching and toning exercises (STRETCH) with education on healthy lifestyle related to brain health (ED). All groups that receive EX and/or DIET will also receive the "Adult Strategies Put Into Real World Environments" (ASPIRE) goal strategy training, with goals focused on exercise and/or diet in order to overcome barriers and increase maintenance of lifestyle changes. All intervention sessions and assessment visits will be conducted online using the Zoom Healthcare platform, and participants will log on using their own devices from home.

ELIGIBILITY:
Inclusion Criteria:

1. 65-80 years old
2. Meet criteria for executive SCD

   1. Answer Yes to both following questions:

      * Do you feel like your memory or thinking is becoming worse?
      * Does this worry you?
   2. ≥1SD above age and sex-based means on any of the sub scales of the Comprehensive Executive Function Inventory (CEFI) - Adult Version, indicative of concerns about executive function.
   3. No objective cognitive impairment as indicated by:

      * A global Clinical Dementia Rating (CDR) of ≤ 0.5
      * A Blind Montreal Cognitive Assessment (MoCA) total score of >17
3. Able to communicate in English
4. Residents of Quebec, Ontario, Manitoba, and Saskatchewan to facilitate concurrent intervention delivery
5. Low physical activity levels (<75min/week of moderate/vigorous physical activity on the Get Active Questionnaire)
6. Screened safe to participate in moderate exercise using the Get Active Questionnaire or physician approval to engage in moderate intensity exercise without in-person supervision
7. Poor diet quality (below Canadian older adults' median intake of fruits, vegetables, nuts and fish, reported using our Diet Screening Questionnaire)
8. Able to participate remotely (i.e., availability of, or ability/willingness to adopt, a computer or tablet alongside high speed internet/data networks)

Exclusion Criteria:

* Dementia, stroke, or other chronic brain disease
* Chemotherapy or radiation to the head/neck in the past year
* Sensory impairments that would impede participation in the intervention or assessments
* Major psychiatric disorder
* Ongoing alcohol or drug abuse that in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
* Contraindications for exercise as determined by the American College of Sports Medicine criteria

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment | 6 months
  Recruitment rate per month
Feasibility: Retention | 6 months
  Percent of consented participants who complete the post-intervention assessment of executive function
Feasibility: Adherence | 6 months
  Percent of study intervention sessions attended by type
Feasiliby: Adherence (diet) | 6 months
  Change in diet quality as assessed with the Eating Pattern Self-Assessment (minimum score 0, maximum score 15; higher scores indicate better diet quality)

SECONDARY OUTCOMES:
Retention by gender | 6 months
  Does retention vary by gender (men, women, other)
Adherence by gender | 6 months
  Does adherence vary by gender (men, women, other)
Executive Function | 6 months
  the primary outcome of a future, large scale trial: an executive function composite derived from Cambridge Brain Sciences on-line assessments, where calculated effect size, variance, and co-variance will inform the sample size for the future, definitive RCT.
Memory | 6 months
  a secondary outcome of a future, large scale trial: memory (Rey Auditory verbal Learning Test [RAVLT] immediate and delayed recall)
Diet | 6 months
  a secondary outcome of a future, large scale trial: diet quality (adherence to the study diet assessed by a study-specific questionnaire [Eating Patterns Self Assessment questionnaire: minimum score 0, maximum score 15; higher scores indicate better diet quality])
Physical Activity | 6 months
  a secondary outcome of a future, large scale trial: physical activity (Physical Activity Scale for the Elderly [PASE], higher scores indicated more physical activity)
Physical Function | 6 months
  a secondary outcome of a future, large scale trial: physical function (assessed using a 5 times sit-to-stand test)
Health-related quality of life | 6 months
  a secondary outcome of a future, large scale trial: Health-related Quality of Life assessed using the SF-36; minimum score 0, maximum score 100, higher scores indicate better quality of life)
Waist Circumference | 6 months
  a secondary outcome of a future, large scale trial: waist circumference
Maintenance of change in executive function | 12 months
  Differences in executive function betwen 6 and 12 months (6 months post-intervention) in an executive function composite derived from Cambridge Brain Sciences on-line assessments
Maintenance of diet quality | 12 months
  Differences in diet quality (as measured by the Eating Patterns Self-Assessment questionnaire: minimum score 0, maximum score 15; higher scores indicate better diet quality) between 6 and 12 months (6 months post-intervention)
Maintenance of physical activity | 12 months
  Differences in physical activity (as measured by the Physical Activity Scale for the Elderly, higher scores indicate greater physical activity) between 6 and 12 months (6 months post-intervention)
Effect modification of executive function by sex | 6 months
  To examine differences in observed effect sizes of executive function (as measured by an executive function composite derived from Cambridge Brain Sciences on-line assessments) vary by sex (male/female)
Effect modification of executive function by gender | 6 months
  To examine differences in observed effect sizes of executive function (as measured by an executive function composite derived from Cambridge Brain Sciences on-line assessments) vary by gender (men, women, other)
Effect modification of physical activity by sex | 12 months
  To examine differences in observed effect for physical activity (as measured by the Physical Activity Scale for the Elderly, higher scores indicate more physical activity) vary by sex (male/female)
Effect modification of physical activity by gender | 12 months
  To examine differences in observed effect for physical activity (as measured by the Physical Activity Scale for the Elderly, higher scores indicate more physical activity) vary by gender (men, women, other)
Effective modification of diet quality by sex | 12 months
  To examine differences in observed effect sizes for diet quality (measured by Eating Patterns Self-Assessment questionnaire; minimum score 0, maximum score 15, higher scores indicate better diet quality) by sex (male/female)
Effective modification of diet quality by gender | 12 months
  To examine differences in observed effect sizes for diet quality (measured by Eating Patterns Self-Assessment questionnaire; minimum score 0, maximum score 15, higher scores indicate better diet quality) by gender (men, women, other)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Middleton, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IDP will be uploaded to an open access data repository. The exact repository has yet to be decided. All data will be de-identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol, analysis plan, and consent forms will become available shortly after ethics approval.
  Clinical study reports will become available after the last data collection and analysis in December 2025. The data will remain on the repository indefinitely.
Access Criteria: Open access

REFERENCES:
- [Derived] Neudorf B, Koblinsky N, Power K, Binns M, Fiocco AJ, Rotenberg S, Marzolini S, Oh P, Thornton J, Ajwani F, Sullivan K, Chevalier S, Russell C, Ferland G, Anderson ND, Middleton LE. Rationale and protocol of the LEAD 2.0 study: a randomized controlled trial assessing the feasibility of a virtually delivered 6-month exercise and nutrition intervention in older adults with subjective cognitive decline (SCD). Pilot Feasibility Stud. 2025 May 10;11(1):64. doi: 10.1186/s40814-025-01626-4. PMID 40349092